CLINICAL TRIAL: NCT06138691
Title: Medication-assisted Psychotherapy: Using Ketamine-enhanced Radically Open Dialectical Behavior Therapy (RO DBT) to Target Neural and Behavioral Mechanisms of Action in Adults With Moderate to Severe Depression
Brief Title: KET-RO Plus RO DBT for Treatment Resistant Depression
Acronym: KET-RO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202212113
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Infusion (Experimental)
  Interventions: Combination Product: Ketamine Infusion plus RO DBT
- Radically Open Dialectical Behavior Therapy (RO DBT) (Experimental)
  Interventions: Combination Product: Ketamine Infusion plus RO DBT

INTERVENTIONS:
Combination Product: Ketamine Infusion plus RO DBT — The participant will receive 4 weeks of 0.5mg/kg intravenous ketamine given over 40 minutes, as is routinely done in ketamine treatment and four months of RO DBT treatment.

SUMMARY:
This pilot study will assess the safety and feasibility of intravenous (IV) ketamine combined with RO DBT in young adults with Treatment-Resistant Depression (TRD). In addition, this study will develop and utilize innovative methodological approaches to demonstrate the feasibility of precision medicine with this type of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-65
* Moderate to severe persistent depression [treatment resistant depression - TRD] (exhibiting 2+ unipolar major depression episodes (non-delusional) with prior treatment non-response to antidepressant or psychosocial treatment
* Treatment-resistant depression: defined as unipolar major depressive disorder, non-delusional (diagnosed by SCID-5, Structured Clinical Interview for the DSM ) that persists despite ≥ 2 adequate antidepressant trials of different classes in the current episode; including at least one evidence-based second-line treatment in the current episode (including serotonin norepinephrine reuptake inhibitors, bupropion, tricyclics, monoamine oxidase inhibitors, or augmentation with an atypical antipsychotic, stimulant, bupropion, lithium, or Triiodothyroinine) higher proportion of OC (over controlled) words endorsed compared to UC (Under controlled) words on the Word Pairs Checklist
* no current or past psychosis
* English speaking
* Able to attend in-person behavioral sessions and ketamine/therapy visits
* Willingness to have RO DBT-A as only psychosocial treatment engaged in (medication treatment may continue-but see below for exclusion)

Exclusion Criteria:

* Outside age range
* Significant neurological condition (i.e., seizure, stroke, severe head injury) or mental retardation (IQ<70)
* Current or recent substance use disorder, actively suicidal or homicidal (e.g., requires hospitalization)
* Use of naltrexone, memantine or medication considered contraindicated with ketamine
* Baseline systolic BP > 150 systolic or 90 diastolic at evaluation. Participants who initially present with elevated blood pressure may be re-assessed; and if needed, referred to their healthcare provider for hypertension management
* Taking more than 2 adequately-dosed oral antidepressants
* Inability to understand, speak and read English sufficiently
* Not be pregnant or at risk of becoming pregnant
* Medical conditions or medication usage that in the judgement of the investigators puts the patient at unreasonable safety risk
* First degree relative with a psychotic diagnosis involving hallucinations, delusions, or disorganized thinking and speech (e.g. schizophrenia, schizoaffective disorder, etc)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Remission from Depression | Approximately 5 months
  Remission defined as Montgomery and Asberg Depression Rating Scale (MADRS) score ≤10. Scale ranges from 0-60 with higher scores indicating higher depression severity.

SECONDARY OUTCOMES:
Visual analogue scale of depressive and anxiety symptoms | Daily following ketamine and therapy sessions during 4 weeks of ketamine-assisted RO DBT
  Asses daily changes in symptoms following ketamine infusions and RODBT sessions
RewP | Approximately 5 months
  The RewP is a neural marker of reward responding and is EEG based. It will examine change id-treatment (Post Ketamine) and post treatment
ERN | Approximately 5 months
  The ERN is a neural marker of error monitoring and is EEG based. It will examine mechanistic change mid-treatment (post ketamine) and post-treatment.
SCS-R and UCLA Loneliness Scale | Approximately 5 months
  The Social Connectedness SCale Revised (SCS-R) and the UCLA loneliness scale measure social connectedness (or lack of) via self-report. They will examine mechanistic change mid-treatment (post ketamine) and post-treatment.

OTHER OUTCOMES:
Temporal Experience of Pleasure Scale (TEPS) | Approximately 5 months
  The TEPS is a self-report behavioral assessment, This measure assesses anticipatory pleasure and consummatory or outcome pleasure of reward responding. It will examine mechanistic change mid-treatment (post ketamine) and post-treatment.
Action and Acceptance Questionnaire (AAQ) | Approximately 5 months
  The AAQ is a self-reported beahvioral measure of psychological ﬂexibility. It will examine mechanistic change mid-treatment (post-ketamine) and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Gilbert, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No